CLINICAL TRIAL: NCT04573972
Title: Using Social Connectedness to Increase Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Principal Investigator, Gretchen Chapman, Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY2019_00000296
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-10

CONDITIONS: Activity, Motor; Social Isolation
Keywords: incentives
MeSH Terms: conditions — Motor Activity; Social Isolation

STUDY DESIGN:
Intervention Model Description: Two group, between-subjects design
Who Masked: Outcomes Assessor
Masking Description: The primary outcome is steps walked, as assessed via the Fitbit app, which is blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular incentive (Active Comparator): During the two-week intervention period, the standard incentive group will earn $2 per day when they meet their step goal, and this reward is earned regardless of whether they walk alone or with others.
  Interventions: Behavioral: Standard Incentive
- Social Incentive (Experimental): During the two-week intervention period, he social incentive group will earn $1 per day when they meet their step goal and an additional $1 if they walk 2,000 steps together with another study participant.
  Interventions: Behavioral: Social Incentive

INTERVENTIONS:
Behavioral: Social Incentive — Receiving half the monetary incentive conditional on meeting a step goal and half the monetary incentive conditional on walking together
  Arms: Social Incentive
Behavioral: Standard Incentive — Receiving the full monetary incentive conditional on meeting a step goal and not conditional on walking together
  Arms: Regular incentive

SUMMARY:
A randomized controlled trial will test the effectiveness of social incentives relative to traditional incentives in promoting walking behavior among college students (N=200). Participants who are rewarded for walking together will be compared to those who are rewarded for walking even when alone. Research participants will download activity tracking apps (Fitbit app and AWARE app) that provide activity and location data. Participants will be consented and then randomized to one of two incentive schemes for walking. Over a 2-week intervention period, the standard incentive group will earn $2 per day when they meet their walking goal regardless of whether they walk alone or with others. The social incentive group will earn $1 per day when they reach their walking goal plus an additional $1 when they walk at least 2000 steps with their walking partner. The incentive scheme will be in place for 2-weeks, preceded by a 1-week baseline period and followed by a 2-week follow-up period.

DETAILED DESCRIPTION:
The objective of the study is to test whether social incentives that encourage physical activity with another person are more effective than incentives for individual exercise. Physical inactivity and social isolation are growing epidemics linked to increased morbidity and mortality particularly among aging Americans. This research aims to address both problems by encouraging co-productive physical activities among college students. Co-productive physical activity mean anything involving physical activity that two people can do together, e.g., walking their dogs or shopping together. Additionally, in light of the COVID-19 pandemic, walking together in this study means either walking while communicating digitally or over the phone, or by physically walking together while wearing a mask, staying 6 feet apart, and following the recommendations from health professionals. A small randomized controlled trial will test the effectiveness of social incentives relative to traditional incentives in promoting walking behavior. Participants who are rewarded for walking together will be compared to those who are rewarded for walking even when alone. The results will indicate whether social incentives are more motivating than traditional incentives for walking behavior.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Able to read and understand English-language surveys
* Own either iPhone or Android smartphones
* Willing to carry the smart phone during the study period and to respond to daily texts or emails from the study team
* Registered for the study as a dyad (friend pairs), with one member of the dyad a Carnegie Mellon University student

Exclusion Criteria:

• Contraindications for increased physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2021-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GRETCHEN B CHAPMAN, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified data will be shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note: all number shown here represent individual participants (not dyads).
Period: Overall Study
Arm/Group | Regular Incentive | Social Incentive
Started | 88 | 84
Completed | 56 | 70
Not Completed | 32 | 14
Not completed — Dyad partner did not join study or did not walk >0 steps | 32 | 14

BASELINE CHARACTERISTICS:
Population: Note: numbers indicate individual participants, not dyads.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regular Incentive | Social Incentive | Total
Number analyzed (Participants) | 56 | 70 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Following our pre-registration, we omitted participants from analysis if the participant's dyad partner did not complete enrollment in the study, if the participant did not have at least 1 baseline day where >0 steps were recorded, or if the participant's dyad partner did not have at least 1 baseline day where >0 steps were recorded.
  years | 21.77 (8.34) | 20.16 (5.67) | 20.87 (7.00)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: female | 35 | 44 | 79
  Gender: male | 21 | 20 | 41
  Gender: other | 0 | 5 | 5
  Gender: prefer not to answer | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 51 | 68 | 119
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 31 | 48 | 79
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 19 | 14 | 33
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Steps Walked From Baseline Period (Week 1) to Intervention Period (Weeks 2 and 3)
Description: Change in mean daily steps walked from baseline (week 1) to intervention period (weeks 2 and 3), as recorded on the FitBit app
Time Frame: week 2-3
Population: Numbers refer to individuals (not dyads).
Measure: Least Squares Mean (Standard Deviation); unit: steps per day
Arm/Group | Regular Incentive | Social Incentive
Number analyzed (Participants) | 56 | 70
steps per day | 483.95 (324.64) | 283.77 (344.89)

2. Primary Outcome: Change in Mean Daily Steps Walked From Baseline Period (Week 1) to Follow-up Period (Weeks 4-5)
Description: Change in mean daily steps walked from baseline to follow-up period, as recorded on the FitBit app
Time Frame: week 4-5
Population: Numbers refer to individuals (not dyads).
Measure: Least Squares Mean (Standard Deviation); unit: steps per day
Arm/Group | Regular Incentive | Social Incentive
Number analyzed (Participants) | 56 | 70
steps per day | 7.33 (271.25) | 159.76 (240.34)

3. Primary Outcome: Mean Number of Days Met Daily Step Goal During Intervention Period (Weeks 2-3) Minus Mean Number of Days Met Same Level of Walking in Baseline Period (Week 1)
Description: Mean number of days when an individual's number of steps walked was at or above daily goal during the intervention period (weeks 2 & 3) minus the mean number of days the individual's number of step's walking was at or above that same level during the baseline period (week 1)
Time Frame: week 2-3
Population: Numbers refer to individuals (not dyads).
Measure: Least Squares Mean (Standard Deviation); unit: days
Arm/Group | Regular Incentive | Social Incentive
Number analyzed (Participants) | 56 | 70
days | 0.03 (0.05) | 0.01 (0.05)

4. Primary Outcome: Mean Number of Days Met Daily Step Goal During Follow-up Period (Weeks 4-5) Minus Mean Number of Days Met Same Level of Walking in Baseline Period (Week 1)
Description: Mean number of days when an individual's number of steps walked was at or above daily goal during the follow-up period (weeks 4 & 5) minus the mean number of days the individual's number of step's walking was at or above that same level during the baseline period (week 1)
Time Frame: week 4-5
Population: Numbers refer to individuals (not dyads).
Measure: Least Squares Mean (Standard Deviation); unit: days
Arm/Group | Regular Incentive | Social Incentive
Number analyzed (Participants) | 56 | 70
days | -0.04 (0.04) | -0.02 (0.05)

5. Primary Outcome: Change in Score on University of California Los Angeles (UCLA) Loneliness Scale (Survey Measure)
Description: 20-item scale measuring subjective feelings of loneliness and social isolation. Minimum score = 0; maximum score = 60; higher scores indicate more loneliness. We computed the difference in score from baseline (beginning of week 1) to end of study (end of week 5).
Time Frame: week 5
Population: Numbers refer to individuals (not dyads).
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regular Incentive | Social Incentive
Number analyzed (Participants) | 56 | 70
score on a scale | -0.01 (0.08) | 0.02 (0.09)

6. Secondary Outcome: Fraction of Days Participant Walked Together With Partner (Self Report) During Intervention Period (Weeks 2-3)
Description: Fraction of days with self report of walking at least 2,000 steps with another participant during intervention period (weeks 2-3)
Time Frame: week 2-3
Population: Numbers refer to individuals (not dyads).
Measure: Least Squares Mean (Standard Error); unit: proportion of days
Arm/Group | Regular Incentive | Social Incentive
Number analyzed (Participants) | 51 | 67
proportion of days | 0.138 (0.065) | 0.535 (0.070)

7. Secondary Outcome: Fraction of Days Participant Walked Together With Partner (Self Report) During Follow-up Period (Weeks 4-5)
Description: Fraction of days with self report of walking at least 2,000 steps with another participant during follow-up period (weeks 3-5)
Time Frame: week 4-5
Population: Numbers refer to individuals (not dyads).
Measure: Least Squares Mean (Standard Error); unit: proportion of days
Arm/Group | Regular Incentive | Social Incentive
Number analyzed (Participants) | 51 | 64
proportion of days | 0.135 (0.077) | 0.408 (0.086)

8. Secondary Outcome: Proportion of Days Participant Walked Together With Partner (Coded)
Description: A machine learning (ML) algorithm will compare the walking records from the Aware app of each dyad of participants and assess whether they walked together on each day
Time Frame: week 2-3
Population: Participants with step data available for algorithm estimate
Measure: Mean (Standard Error); unit: proportion of days walked together
Arm/Group | Regular Incentive | Social Incentive
Number analyzed (Participants) | 34 | 30
proportion of days walked together | 0.5564 (0.06213) | 0.7091 (0.06306)

9. Secondary Outcome: Proportion of Days Participant Walked Together With Partner (Coded)
Description: as for outcome 8
Time Frame: week 4-5
Population: Participants with step data available for algorithm estimate
Measure: Mean (Standard Error); unit: proportion of days walked together
Arm/Group | Regular Incentive | Social Incentive
Number analyzed (Participants) | 30 | 24
proportion of days walked together | 0.5444 (0.07536) | 0.6583 (0.08425)

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Definitions do not differ
  Note: Numbers below indicate individuals (not dyads) The number of "at risk" individuals includes all individuals who started the study flow, even those that did not meet inclusion criteria and did no receive any intervention.
Arm/Group | Regular Incentive | Social Incentive
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/84
Other Adverse Events (participants affected / at risk) | 0/88 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT04573972/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT04573972/SAP_001.pdf